CLINICAL TRIAL: NCT05588102
Title: Research on Standardized Electronic Cognitive Training Technique in Early Stage of Senile Depression With Cognitive Impairment
Brief Title: Electronic Training of Elderly Depression With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Qinge Zhang, prof, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z191100006619061
Record Dates: First submitted 2022-08-17; First posted 2022-10-20 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Geriatric Depression; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Paroxetine; Fluvoxamine; Sertraline; Citalopram; Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective Serotonin Reuptake Inhibitor（SSRIs）combined with Electronic cognitive training (Experimental): SSRIs（Fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, escitalopram）combined with Electronic cognitive training (60min, once a day)
  Interventions: Drug: Selective Serotonin Reuptake Inhibitor（SSRIs，Fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, escitalopram）
- SSRIs antidepressants combined with blank control Electronic training for 52 weeks (Placebo Comparator): SSRIs drug treatment （Fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, escitalopram）combined with the blank control Electronic training(subjects were allowed to use electronic products to browse the web and watch the news for 1 hours every day)
  Interventions: Drug: Selective Serotonin Reuptake Inhibitor（SSRIs，Fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, escitalopram）

INTERVENTIONS:
Drug: Selective Serotonin Reuptake Inhibitor（SSRIs，Fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, escitalopram） — Subjects in the intervention group received SSRIs antidepressants combined with Electronic cognitive training based on mobile phone platform for 52 weeks (once a day, 60min each time)
  Other Names: Electronic cognitive training

SUMMARY:
late-life depression (LLD) is the most common mental illness in the elderly. Due to the increasing prevalence of population aging, it has become one of the important factors affecting the quality of life of the elderly. 50-70% of elderly patients with depression are accompanied by different degrees of cognitive impairment.

DETAILED DESCRIPTION:
Elderly patients with depression with cognitive impairment have a greater risk of dementia conversion, a worse prognosis and a higher recurrence rate. Therefore, it is urgent to provide evidence-based early intervention strategies for geriatric depression with cognitive impairment. At present, domestic and foreign guidelines do not provide clear and effective treatment plans for elderly patients with depression with cognitive impairment, and clinical research and practice also lack evidence-based treatment methods. Selective Serotonin Reuptake Inhibitors (SSRIs), the most commonly used antidepressants, do not significantly improve the cognitive impairment of elderly patients with depression, and may even aggravate the cognitive impairment of elderly patients with depression. The overall efficacy and tolerability of drug therapy in elderly patients with depression and cognitive impairment are poor. Studies have confirmed that Cognitive training can significantly improve the overall Cognitive function and multiple Cognitive domains of healthy elderly people, patients with Mild Cognitive Impairment (MCI) and Alzheimer's disease (AD). Previous studies have also preliminarily confirmed the cognitive improvement effect of cognitive training on elderly patients with depression, which provides a new idea for clinical diagnosis and treatment. Therefore, based on the urgent clinical needs and preliminary work, the development and clinical validation of a set of standardized cognitive training methods suitable for elderly patients with depression and cognitive impairment will be conducive to improve the overall efficacy of elderly patients with depression, improve the prognosis of patients, and save health resources.

ELIGIBILITY:
Inclusion Criteria:

1. The patients and their family members signed the written informed consent
2. Age ≥60 years old
3. Meet the diagnostic criteria for single or recurrent major depressive disorder in the diagnostic and Statistical Manual of mental disorders Fourth Edition (DSM-V)
4. Currently in the acute phase, HAMD-17 total score at baseline ≥ 18 points
5. There are symptoms of cognitive impairment, Montreal Cognitive Assessment scale (Montreal Cognitive Assessment scale, MoCA) <26 points
6. Education level above primary school.

Exclusion Criteria:

1. Patients with history of epilepsy or coronary heart disease or other serious unstable physical diseases
2. Participated in another intervention clinical study in the past 1 month
3. The following mental diseases have been or are currently diagnosed by DSM-V: organic mental disorder, Alzheimer's disease, secondary dementia caused by other causes, schizophrenia, schizophrenic affective disorder, bipolar disorder, delusional disorder, undefined mental disease, patients with drug abuse history, including alcohol and active drug abuse in the past 12 months, except nicotine
4. He has been taking antidepressants, mental retardants and other psychiatric drugs for the past 2 weeks
5. Severe aphasia, visual and hearing impairment, etc. unable to complete the scale evaluation

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
At the end of the 12th week of treatment, the change value of ADAS-Cog score of subjects in the two groups compared with baseline | 12 week
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) was developed in the 1980s to assess the level of cognitive dysfunction in Alzheimer's disease.The score of the scale is about 0-75 points, and the higher the score, the cognitive function decreases significantly

SECONDARY OUTCOMES:
At each follow-up point, the change value of ADAS cog scale score of subjects in the two groups compared with baseline; | 52week
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) was developed in the 1980s to assess the level of cognitive dysfunction in Alzheimer's disease.The score of the scale is about 0-75 points, and the higher the score, the cognitive function decreases significantly.
At each follow-up point, the change value of HAMD-17 scale score of subjects in the two groups compared with baseline; | 52week
  17-Item Hamilton Rating Scale for Depression (HAMD-17)， Mild depression: HAMD-17 scores > 7 points, ≤ 17 points; Moderate depression: HAMD 17 scores > 17 points, ≤ 24 points;Severe depression: HAMD 17 scores > 24 points.
At each follow-up point, the change value of HAMA scale score of subjects in the two groups compared with baseline; | 52week
  Hamilton Anxiety Scale (HAMA) is used to assess the anxiety level of patients. The 14 item cutoff value of HAMA is 14 points. The higher the score, the more serious the anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Qinge Zhang, PhD, Study Chair — Beijing Anding Hospital Affiliated to Capital Medical University
Locations (1):
- Beijing Anding Hospital Affiliated to Capital Medical University, Beijing, China

REFERENCES:
- [Background] Mulsant BH, Ganguli M. Epidemiology and diagnosis of depression in late life. J Clin Psychiatry. 1999;60 Suppl 20:9-15. PMID 10513852
- [Background] Horackova K, Kopecek M, Machu V, Kagstrom A, Aarsland D, Motlova LB, Cermakova P. Prevalence of late-life depression and gap in mental health service use across European regions. Eur Psychiatry. 2019 Apr;57:19-25. doi: 10.1016/j.eurpsy.2018.12.002. Epub 2019 Jan 15. PMID 30658276
- [Background] Goncalves-Pereira M, Prina AM, Cardoso AM, da Silva JA, Prince M, Xavier M; 10/66 Workgroup in Portugal. The prevalence of late-life depression in a Portuguese community sample: A 10/66 Dementia Research Group study. J Affect Disord. 2019 Mar 1;246:674-681. doi: 10.1016/j.jad.2018.12.067. Epub 2018 Dec 21. PMID 30611911
- [Background] Wang F, Zhang QE, Zhang L, Ng CH, Ungvari GS, Yuan Z, Zhang J, Zhang L, Xiang YT. Prevalence of major depressive disorder in older adults in China: A systematic review and meta-analysis. J Affect Disord. 2018 Dec 1;241:297-304. doi: 10.1016/j.jad.2018.07.061. Epub 2018 Jul 27. PMID 30142588
- [Result] Buchtemann D, Luppa M, Bramesfeld A, Riedel-Heller S. Incidence of late-life depression: a systematic review. J Affect Disord. 2012 Dec 15;142(1-3):172-9. doi: 10.1016/j.jad.2012.05.010. Epub 2012 Aug 30. PMID 22940498
- [Derived] Wang X, Zhou J, Zhu K, Wang Y, Ma X, Ren L, Guo C, Zhang Z, Lu P, Zhang Q. Efficacy and safety of Neurocognitive Adaptive Training for Depression combined with SSRIs for treating cognitive impairment among patients with late-life depression: a 12-week, randomized controlled study. BMC Psychiatry. 2024 Nov 25;24(1):848. doi: 10.1186/s12888-024-06276-z. PMID 39587504

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT05588102/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT05588102/ICF_001.pdf